CLINICAL TRIAL: NCT02569619
Title: Evaluation of an Intervention to Promote Physical Activity in Outpatients With Mental Disorders: Motivational Determinants of Adherence, Effect on Cognitive Determinants of Physical Activity, Physical Activity, Sitting Time and Clinical Symptoms
Brief Title: Evaluation of an Intervention to Promote Physical Activity in Outpatients With Mental Disorders
Acronym: GAF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Moritz Petzold, Dipl.Psych. Moritz Petzold, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAF-1
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Mental Disorders
Keywords: Physical Activity; Mental Health; Physical Exercise; Mental disorder; Promotion
MeSH Terms: conditions — Mental Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity Intervention (Experimental): The activity intervention is MoVo-LISA (Göhner & Fuchs, 2007). A psychological program with two group sessions of 90 minutes and one one-on-one session of about 15 minutes. The patients develop aims for their health, ideas, how to reach these aims through physical activity and make detailed plans, how to implement activity in their everyday routine. Difficulties and barriers are discussed.
  Interventions: Behavioral: Activity Intervention
- Healthy Diet Intervention (Active Comparator): The healthy diet intervention is a modification of MoVo-LISA. A psychological program with two group sessions of 90 minutes and one one-on-one session of about 15 minutes. The patients develop aims for their health, ideas, how to reach these aims through a healthy diet and make detailed plans, how to implement a healthy diet in their everyday routine. Difficulties and barriers are discussed.
  Interventions: Behavioral: Healthy Diet Intervention

INTERVENTIONS:
Behavioral: Activity Intervention
  Arms: Activity Intervention
Behavioral: Healthy Diet Intervention
  Arms: Healthy Diet Intervention

SUMMARY:
The purpose of this study is to determine if a manualised intervention to promote physical activity (MoVo-LISA) is effective to help psychiatric outpatients to increase their level of everyday physical activity.

DETAILED DESCRIPTION:
The Intervention program MoVo-LISA is a psychological intervention that should help participants to increase their level of physical activity for a healthy lifestyle.It contains three sessions (2 group,1 one on one) in the course of two weeks. The intervention focuses on planning and barrier management.

Participants develop activity ideas, goals and plans that enable them to integrate physical activity in their everyday routine and how to shield their motivation against barriers and difficulties.The intervention has proven to be effective with patients with pain disorders in rehabilitation.

This study examines if the intervention if effective for psychiatric outpatients as well. The intervention is compared to an active control group that receives a similar program that is focusing on a healthy diet.

Participants are recruited in the outpatient departements of three hospitals in Berlin and Brandenburg (Charité Universitätsmedizin Berlin - Departement of Psychiatry and Psychotherapy; St. Hewdig Hospital Berlin - Departement of Psychiatry; Oberhavel Hospital Brandenburg, Departement of Psychiatry) and at local psychiatrists in Berlin. Individuals are recruited by posters and flyers in the waiting areas areas or by information of their doctor. Patients can contact the researcher and are, after checked for eligibility, invited to an information event, where they get detailed information on the program and the study. After the information event, participants give written informed consent.

The intervention takes place in the outpatient departements of the three hospitals.

Clinical information about diagnoses, medication and functioning is obtained by their doctors by mail after the patients released them from confidentiality.

The study is an explorative approach to test if the program is suited for psychiatric patients. A sample size of 50 participants that complete the program is planned.

All data is collected pseudonymised to protect the identity of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of Age
* Patients in one of the psychiatric outpatients or at an local psychiatrist in Berlin
* Mental illness (ICD-10: F1-F4)
* No contraindications for physical activity
* Able to understand german language

Exclusion Criteria:

* Contraindications to physical activity
* Acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in physical activity - objective | From baseline (T1) to 3 month after the intervention (T3)
  Physical activity is objectively measured using accelerometry (ActiGraph GT1M)
Change in physical activity - subjective | From baseline (T1) to 3 month after the intervention (T3)
  Physical activity is subjectively measured with the International Physical Activity Questionaire (IPAQ)

SECONDARY OUTCOMES:
Change in self-efficacy | From baseline (T1) to 1 week after the intervention (T2)
  Self-efficacy is measured using two likert scaled items
Change in intention for physical activity | From baseline (T1) to 1 week after the intervention (T2)
  Intention for physical activity is measured using two likert scaled items
Change in self concordance of the motivation for physical activity | From baseline (T1) to 1 week after the intervention (T2)
  Self concordance of the motivation for physical activity is measured using the "Sport- und bewegungsbezogene Selbstkonkordanz Skala", which consists of 12 likert scaled items
Change in outcome expectancies for physical activity | From baseline (T1) to 1 week after the intervention (T2)
  Outcome expectancies for physical activity are measured using 6 likert scaled items
Change in planning for physical activity | From baseline (T1) to 1 week after the intervention (T2)
  Planning for physical activity is measured using 4 likert scaled items
Change in barrier planning for physical activity | From baseline (T1) to 1 week after the intervention (T2)
  Barrier planning for physical activity is measured using 4 likert scaled items
Change in psychopathological symptoms | From baseline (T1) to 3 month after the intervention (T3)
  Psychopathological symptoms are measured by the Symptom Checklist 27 (SCL-27)
Change in health-related quality of life | From baseline (T1) to 3 month after the intervention (T3)
  Health-related quality of life is measured using the Sort-Form Health Questionnaire 12 (SF-12)
Change in dietary behavior | From baseline (T1) to 3 month after the intervention (T3)
  Dietary behavior is measured using the Food Frequency Questionnaire (FEL)
Change in consumption of portions of fruit and vegetable per day | From baseline (T1) to 3 month after the intervention (T3)
  Consumption of fruit and vegetable is measured using two items asking for the number of portions of fruit and vegetable that are consumed on a regular day (a portion is defined as a hand full). Consumption of fruit and vegetable is then added to check if the WHO recommendation of "5 a day" is met

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof., Study Director — Charité Universitätsmedizin Berlin - Departement of Psychiatry and Psychotherapy; Moritz B Petzold, Dipl.Psych., Principal Investigator — Charité Universitätsmedizin Berlin - Departement of Psychiatry and Psychotherapy
Locations (1):
- Charité Universitätsmedizin Berlin - Departement of Psychiatry, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Hardt J, Gerbershagen HU. Cross-validation of the SCL-27: a short psychometric screening instrument for chronic pain patients. Eur J Pain. 2001;5(2):187-97. doi: 10.1053/eujp.2001.0231. PMID 11465984
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Winkler G, Doring A. Validation of a short qualitative food frequency list used in several German large scale surveys. Z Ernahrungswiss. 1998 Sep;37(3):234-41. doi: 10.1007/pl00007377. PMID 9800314
- See also: Information on the MoVo-model and intervention — http://www.sport.uni-freiburg.de/institut/Arbeitsbereiche/psychologie/psych_proj/konz